CLINICAL TRIAL: NCT01234922
Title: A Phase II Study of the Effect of ACE Inhibitors on Pro-Angiogenic Hormones in Cancer Patients With Hypertension
Brief Title: Benazepril Hydrochloride, Lisinopril, Ramipril, or Losartan Potassium in Treating Hypertension in Patients With Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00014933; NCI-2010-02043 (Other: CTRP); IRB00014933 (Other: WFUHS IRB); CCCWFU 98710 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Hypertension; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Hypertension | interventions — Lisinopril; Losartan; benazepril; Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm I (Experimental): Patients receive oral benazepril hydrochloride once daily on days 1-7.
  Interventions: Other: laboratory biomarker analysis; Drug: benazepril hydrochloride
- Arm II (Experimental): Patients receive oral lisinopril once daily on days 1-7.
  Interventions: Drug: lisinopril; Other: laboratory biomarker analysis
- Arm III (Experimental): Patients receive oral ramipril twice daily on days 1-7.
  Interventions: Other: laboratory biomarker analysis; Drug: ramipril
- Arm IV (Experimental): Patients receive oral losartan potassium once daily on days 1-7.
  Interventions: Drug: losartan potassium; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lisinopril — Given orally
  Other Names: Prinivil; Zestril
  Arms: Arm II
Drug: losartan potassium — Given orally
  Other Names: Cozaar
  Arms: Arm IV
Other: laboratory biomarker analysis — Correlative studies
Drug: benazepril hydrochloride — Given orally
  Other Names: benazepril HCl; CGS14824A; Lotensin
  Arms: Arm I
Drug: ramipril — Given orally
  Other Names: Altace
  Arms: Arm III

SUMMARY:
RATIONALE: Benazepril hydrochloride, lisinopril, ramipril, and losartan potassium may help lower blood pressure.

PURPOSE: This phase II trial is studying how well benazepril hydrochloride, lisinopril, ramipril, or losartan potassium works in treating hypertension in patients with solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine which drug has the greatest effect on Ang-(1-7) levels in cancer patients with hypertension.

SECONDARY OBJECTIVES:

I. To determine the effect of these drugs on levels of Ang II, VEGF, PlGF, and ACE in the same patients.

OUTLINE: Patients are randomized to 1 of 4 treatment arms.

* ARM I: Patients receive oral benazepril hydrochloride once daily on days 1-7.
* ARM II: Patients receive oral lisinopril once daily on days 1-7.
* ARM III: Patients receive oral ramipril twice daily on days 1-7.
* ARM IV: Patients receive oral losartan potassium once daily on days 1-7. In all arms, treatment continues in the absence of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed solid tumor malignancy AND hypertension, defined as a systolic pressure > 130 OR a diastolic pressure > 80
* Patients cannot be on active chemotherapy or radiation therapy; start of treatment with ACE-I or ARB must occur at least four weeks after the last dose of chemotherapy or radiation therapy
* Creatinine < 2.5
* Potassium < ULN
* Ability to understand and the willingness to sign a written informed consent document
* HIV positive patients are eligible to participate in this study

Exclusion Criteria:

* Patients who are pregnant or nursing due to significant risk to the fetus/infant
* Patients who are unable to take oral medications
* Patients who are currently taking an ACE-Inhibitor or ARB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Petty, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol was closed early due to slow accrual
Period: Overall Study
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Started | 1 | 1 | 2 | 2
Completed | 1 | 1 | 2 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Arm III | Arm IV | Total
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 2 | 1 | 4
  >=65 years | 0 | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (0) | 68.8 (0) | 62.2 (1.45) | 65.5 (6.15) | 61.7 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 2 | 2
  Male | 1 | 1 | 2 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 2 | 2 | 6
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Changes in Ang1-7 Levels Among Patients After ACE-I/ARB Treatment Measured in Picogram/Milliliter
Time Frame: 7 days post-baseline
Measure: Mean (Standard Deviation); unit: Picogram/milliliter
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 1 | 1 | 2 | 2
Picogram/milliliter | 13.25 (0) | 33.67 (0) | 6.685 (10.815) | 5.045 (5.275)

2. Secondary Outcome: Change in Ang II, VEGF, PlGF, and ACE Levels
Time Frame: 1 week
Population: Data were not analyzed due to insufficient accrual to the study and lack of statistical power.
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 7 days after dosing
Arm/Group | Arm I | Arm II | Arm III | Arm IV
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/2 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=1) | Arm II (N=1) | Arm III (N=2) | Arm IV (N=2)
Hemoglobin (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hyperglycemia (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain, Chest (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
lymphopenia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vomitting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes